CLINICAL TRIAL: NCT03195673
Title: A Pilot Study Assessing the Safety and Efficacy of Low Dosage of Terazosin in Subjects Undergoing Carotid Artery Stenting
Brief Title: Safety and Efficacy of Low Dosage of Terazosin in Subjects Undergoing Carotid Artery Stenting
Acronym: TZ-CAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: The Luhe Teaching Hospital of the Capital Medical University (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TZ-CAS
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid artery stenting; Silent embolism; Terazosin
MeSH Terms: conditions — Carotid Stenosis | interventions — Terazosin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TZ group (Experimental): Treatment:Patients in this group received standard medical therapy and Terazosin (TZ) treatment.
  Drug: TZ 0.5mg once a day for 3-7 days before carotid artery stenting to 30 days later.
  Procedure: Carotid Artery Stenting
  Interventions: Drug: Terazosin; Procedure: Carotid artery stenting
- control group (Other): Treatment: Patients in this group received standard medical therapy alone. Procedure: Carotid Artery Stenting
  Interventions: Procedure: Carotid artery stenting

INTERVENTIONS:
Drug: Terazosin — TZ 0.5mg once a day for 3-7 days before carotid artery stenting to 30 days later.
  Other Names: TZ
  Arms: TZ group
Procedure: Carotid artery stenting — Carotid artery stenting is an alternative treatment of carotid artery stenosis, which would be performed by experienced neuroradiologist according to the latest guideline from American Heart Association and American Stroke Association.
  Other Names: CAS

SUMMARY:
The purpose of this study is to assess the safety and efficacy of low dosage of Terazosin in Carotid Artery Stenting

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic or asymptomatic carotid artery stenosis. In symptomatic patients the degree of stenosis should more than 50% (Based on NASCET Criteria), in asymptomatic patients the degree of stenosis should more than 70% (Based on NASCET Criteria);
2. Tolerance to any of the study medications, including TZ, clopidogrel, aspirin and statins;
3. Hypertensive patients with or without oral antihypertensive drugs
4. Can cooperate with and complete brain MRI examination;
5. Stable vital signs, cardiopulmonary, liver and kidney function was no obvious abnormalities;
6. Has a negative pregnancy test within 7 days before randomization and no childbearing potential;
7. Stable vital sign, normal renal and hepatic functions;
8. Informed consent.

Exclusion Criteria:

1. Evolving stroke;
2. Hemorrhagic tendency；
3. Severe dementia or Prior major ipsilateral stroke, if likely to confound study endpoints;
4. Chronic atrial fibrillation or any other Cardiogenic emboli source disease;
5. Myocardial infarction within previous 30 days;
6. Spontaneous Intracerebral Hemorrhage within the past 180 days, Hemorrhagic conversion of an ischemic stroke within the past 60 days or recent (<7 days) large area cerebral infarction has a hemorrhagic conversion tendence;
7. Any conditions that hampers proper angiographic assessment or makes percutaneous arterial access unsafe;
8. High risk candidates of CAS defined as the Carotid Revascularization Endarterectomy vs. Stenting Trial (CREST);
9. Thiazides taken within 14 days before randomization;
10. Participating in any other clinical trial that has not completed the required protocol follow-up period;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Participants who got New DWI Lesions (MRI) | Within 48 hours after carotid artery stenting
  Patients who got new ischemic lesions as defined by DWI MRI within 48 hours after carotid artery stenting

SECONDARY OUTCOMES:
Number of New DWI Lesions (MRI) | Within 48 hours after carotid artery stenting
  Number of new ischemic lesions as defined by DWI MRI within 48 hours after carotid artery stenting
Volume of New DWI Lesions (MRI) | Within 48 hours after carotid artery stenting
  Volume of new ischemic lesions as defined by DWI MRI within 48 hours after carotid artery stenting
Number of patients with New DWI Lesions (MRI) diameter greater than 5mm | Within 48 hours after carotid artery stenting
  Patients who got new ischemic lesions diameter greater than 5mm as defined by DWI MRI within 48 hours carotid artery stenting
Number of Patients with Cerebrovascular Events, Cardiovascular Events or Death. | From baseline to 30 days after treatment
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage and hyperperfusion syndrome. Cardiovascular events included angina and myocardial infarction. Death included any reason caused death.
Laboratory Examination | Before and 24 hours after carotid artery stenting
  Laboratory Examination before and post-treatment
Number of Patients underwent hypertensive treatment due to post-procedure hypotention | 0-7 days or discharge which comes early
  Number of Patients underwent hypertensive treatment due to post-procedure hypotention
Number of Patients with Any Side Events | From baseline to 30 days after treatment
  Any side events caused by TZ, regular treatment or CAS
Mortality | From baseline to 30 days after treatment
  Any cause of death

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The Luhe Teaching Hospital of the Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes